CLINICAL TRIAL: NCT04803695
Title: Role of Pseudomonas Aeruginosa Biofilms in Exacerbations in Patients With Bronchiectasis With and Without Chronic Obstructive Pulmonary Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: ISCIII (Unknown)
Responsible Party: Sponsor
Other Study IDs: v.11 27/02/18
Record Dates: First submitted 2021-03-11; First posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Bronchiectasis; Microbial Colonization; Pseudomonas Aeruginosa; Biofilm
MeSH Terms: conditions — Bronchiectasis; Communicable Diseases; Pseudomonas Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sputum Serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Microbial biofilm diagnose — Usage of new microbiological methods for biofilm detection

SUMMARY:
Exacerbations, in particular during chronic Pseudomonas aeruginosa (PA) infection, are very important in the prognosis of patients with non-cystic fibrosis bronchiectasis (BE). In Cystic Fibrosis patients, PA biofilms are associated with chronic respiratory infections and are the primary cause of their increased morbidity and mortality. However, the presence and role in exacerbations of PA biofilms, microbiome dysbiosis and inflammatory biomarkers has not been studied in depth in BE patients. Our aim is to determine the association between PA chronic infection and its biofilms with the number of exacerbations in the next year (primary outcome), time until next exacerbation, quality of life, FEV1 and inflammatory biomarkers (secondary outcomes) in BE patients with or without chronic obstructive pulmonary disease (COPD). The investigators will include and follow up during 12 months post study inclusion, 48 patients with BE and 48 with BE-COPD, with a positive sputum culture of PA. During stability and follow up (and in each exacerbation) The investigators will collect 4 sputum, 4 serum samples, perform spirometry, and quality of life tests every three months. For the biomarkers subproject, 4 additional serum samples will be collected at: exacerbation, 3-5 days after treatment, at 30 days and three months post-exacerbation. Biomarkers will be measured by commercial kits and Luminex. The investigators will quantify PA colony forming units (CFU)/mL, their resistance pattern, their mutation frequency and isolate mucoid and non-mucoid colonies. In each sputum, the investigators will analyze by Confocal Laser Scanning Microscopy (CLSM) and Fluorescent in situ Hybridizatrion (FISH) PA biofilms, their size, bacterial density and their in situ growth rate. Specific serum antibodies against PA will be determined through Crossed Immunoelectrophoresis. In addition, the investigators will indentify potential respiratory microbiome and gene expression patterns predictive for exacerbations, or with a protective role against chronic PA infection, as well as their association with biofilms. Microbiome analysis will be performed through the Illumina Miseq platform. Finally, the investigators will explore the antimicrobial activity of novel combinations of antibiotics against PA, both in in vitro planktonic cultures and in a biofilm model, and will include testing of antibiotic-containing alginate nanoparticles.

DETAILED DESCRIPTION:
This project will study the association between chronic PA infection in the airways and the formation of biofilms in the following patient populations: 1-bronchiectasis not associated with cystic fibrosis (BQ) and 2-bronchiectasis with chronic obstructive pulmonary disease (BQ-EPOC). The primary objective is to determine the association between chronic infection by PA, presence of biofilms of PA and the worst evolution of the disease measured mainly by the number of exacerbations per year (primary outcome) days until the next exacerbation, quality of Life and Forced Expiratory Volume (FEV1), and inflammatory biomarkers (secondary outcomes). For this, these parameters will be compared in patients with chronic infection by PA and with the presence of biofilms of PA in the sputum (identified by FISH-CLSM) vs those with PA without chronic infection and without biofilms (control negative) in each study population (BE and BE-COPD). The investigators will analyze, to the recruitment and sequentially (3 determinations), various aspects of the biofilms that are detailed in the methodology. In addition, by comparing the microbiome before, during and after each exacerbation, the investigators will try to identify those microbial patterns that entail a higher risk of exacerbation, those with a protective role against chronic PA infection and its relationship with biofilms.

The diagnosis of biofilms is not yet routinely implemented in clinical practice for Chronic Obstructive Pulmonary Disease (COPD) and NonCF Bronchiectasis (BE) infections. The first guidelines for the diagnosis and treatment of biofilm infections were published in 2015 and included many biofilm-associated infections, but not COPD or BE. There are in fact very few studies on the presence of PA biofilms in these populations and on their potential role in exacerbations. However, there is sound scientific evidence that PA biofilms are associated with chronic respiratory infections in Cystic Fibrosis (CF) patients, and are the primary cause of their increased morbidity and mortality. It has been reported that during chronic PA lung infection in CF, PA adapts to different niches in the lungs. Both mucoid (biofilms) and non-mucoid (planktonic) bacteria are present in sputum. Cells with higher mutation rate develop multi-resistance to many antibiotics and their in situ growth rate is lower, since bacteria decrease their metabolism conditioned by high polymorphonuclear oxygen consumption, As yet, however, none of this has been described in patients with BE; in fact, there are very few studies on the presence of PA biofilms in these populations, and their role in the exacerbations has not been demonstrated. In addition, there is little evidence of the association of the microbiome dysbiosis with chronic colonization by PA and during exacerbations.

Chronic colonization by PA is present in 12-27% of patients with BE and BE-COPD, and entails a worse prognosis (a 3-fold increase in mortality risk) and up to a 7-fold increase in the risk of hospital admission, with an average of one additional exacerbation per patient and per year. In these patients, eradication of PA is difficult, despite the fact that an adequate antimicrobial treatment reduces the bacterial load and the number of exacerbations and improves lung function and quality of life. One of the main challenges in patients with BE is the eradication of PA, especially during the early stages of colonization by this pathogen. In this situation, aggressive antibiotic treatment is recommended. However, this eradication fails in a notable percentage of cases. In addition to the increase in multiresistance in PA, even against quinolones, its ability to produce biofilms and survive in them is one of the reasons for the failed eradication. Although the presence of PA in sputum is a factor of poor prognosis in BE, biofilms have not yet been identified and characterized (i.e., their presence, size, amount of alginate and metabolic status) in sputum of these populations. Recently, the presence of biofilms in bronchoalveolar lavage (BAL) samples has been described by confocal laser scanning microscopy (CLSM) in pediatric patients with BE, even in those samples in which the culture was negative. This finding draws attention to the lack of studies on biofilm in BE and the importance of improving diagnostic tools for detection in respiratory samples, especially in patients with recurrent exacerbations despite antibiotic treatment.

Between 30 and 50% of patients with moderate or severe COPD have BE. Its prevalence increases with the severity of COPD, while 5-10% of patients with BE have COPD. Patients with COPD and BE form a clinical group with its own characteristics (increased sputum production and purulence, greater dyspnea and number of exacerbations), worse prognosis, possible therapeutic implications and higher mortality. Although the causes of exacerbations are not yet well understood, bacterial infections are thought to be involved in approximately one-half of cases PA is one of the most frequent pathogens isolated from these exacerbations and is associated with higher mortality. PA from sputum of chronically infected COPD patients tends to be less cytotoxic and motile and produces more biofilm than PA from blood samples. Therefore, some authors suggest that COPD, BE and CF present similar patterns of infection and evolution. Following this reasoning, our hypothesis is that PA biofilms could be one of the pathogenic mechanisms associated with both the persistence of infections and the frequency and severity of exacerbations in patients with BE (with or without COPD). However, further research using the recommendations of the current guidelines is needed to confirm this hypothesis.

Some authors who have studied microbial dysbiosis in COPD exacerbations have seen that, along with eosinophilic inflammation, it is associated with more severe exacerbations and a greater fall in lung function. Longitudinal studies of the microbiome in the sputum of patients with BE suggest that the management of chronic bronchial infection can be improved with a therapy that is specific for its microbiome, taking into account the burden of the pathogen, the stability of the community, and acute and chronic community responses to antibiotics. However, the fluctuations in the microbiome and its predictive role in the exacerbations of bronchiectasis have not yet been studied in depth. The study of variations in the microbiome before and during the exacerbation could reveal novel therapeutic targets that may have an impact on the management of patients. The results could help to determine the need to administer antimicrobial treatment in patients with negative microbiological cultures during the exacerbation. There is evidence that a balanced oral flora could have a protective role against the colonization of saliva by PA; however, a microbiome pattern with a protective effect on the upper respiratory tract against PA in BE patients and its relationship with PA biofilms has not yet been described.

Simultaneously, systemic biomarkers and inflammatory cytokines determine the potential importance of chronic PA infection and the productions of biofilms. Systemic CRP has been shown to be correlated with higher BE scores such as FACED and BSI. However, there are no longitudinal studies evaluating the intensity and duration of systemic inflammation caused by chronic PA infection.

The spread of antibiotic resistance and increasing prevalence of biofilm-associated infections is driving demand for new means to treat such difficult to eradicate bacterial infections. Recently, the WHO published a list of bacteria for with research on new antibiotics is urgently needed. Drug discovery and development is a tedious, long and costly endeavour that can take hundreds of millions EUR and 10-15 years from the bench discovery to the bedside. Chronic PA infections associated to BE are typically treated with combinations of up to three antimicrobials. Despite periodic courses of multidrug therapy, effective cure for these diseases is below optimal levels. It is clear then that new therapeutic options are needed to improve positive outcomes in these patients. Our approach focuses on the concept of synergy, i.e. identifying synergistic combinations of antibiotics, being together more effective that when used alone. The investigators aim to systematically evaluate the synergistic interactions of currently used antibiotics and explore the introduction of other clinically approved antibiotics. Since their pharmacology and toxicity has been already well documented, any potential synergistic antibiotic combination could progress to clinical trials at fraction of the standard development cost and in much shorter period of time. Along with this, the nanocarrier-mediated delivery strategy has been suggested as a promising approach in treatment of drug resistant infections. Nanotechnology may provide an innovative platform for addressing the challenge of PA chronic infections associated to bronchiectasis, with potential to manage difficult to treat infections involving multidrug-resistant (MDR) bacteria. In particular, polysaccharide (PS)-based nanocarriers are ideal vehicles for encapsulation of antimicrobials and alginate is an ideal carrier for pulmonary administration due to its mucoadhesive properties.

ELIGIBILITY:
Inclusion Criteria:

* BE criteria (with and without COPD)
* Isolation of PA in sputum in the stable phase. * A prospective screening of BQ patients in outpatient consultations will be conducted to prospectively detect those with isolation of PA in the sputum.

Exclusion Criteria:

* CF
* Immunosuppression (primary and secondary, with the exception of cases of IgG deficiency in stable substitution treatment)
* Sarcoidosis
* Tuberculosis, active infection by nontuberculous mycobacteria
* Diffuse interstitial lung disease
* Altered state of consciousness or disability to understand the study and perform the tests provided by it, involving the patient in another intervention study (clinical trials).

  * Patients with CF are excluded because the role of PA biofilms in CF has been extensively studied, as argued in the background of the present proposal and the selected literature. It is also a totally different disease from the one we intend to study, with patients of much younger ages. Finally, this is a very vulnerable population in which it would be very difficult to obtain all the samples sequentially.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 96 BE patients (48 with BE and 48 with BE-COPD), and with positive sputum culture for PA. Follow-up will be performed for 12 months after the first isolation of PA. All patients must sign informed consent before recruitment in the study.
Sampling Method: Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of exacerbations per year | 1 year
  Exacerbations during the follow up

SECONDARY OUTCOMES:
Levels of inflammatory biomarkers during the follow up and in exacerbations | 1 year
  During exacerbation: Samples (plasma and serum) will be extracted on day 1, at 3-5 days of treatment, at 30 days and at 3 months after the exacerbation. They will be coded and they will be frozen until analysis.
  Stable phase: Samples (plasma and serum) will be extracted, coded and frozen until analysis. Determination of cytokines:
  IL-17, IL-6, IL-8, TNFa, IL-1b by commercial kits and Luminex.

CONTACTS AND LOCATIONS:
Overall Officials: Fernández-Barat Laia, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hoiby N, Bjarnsholt T, Moser C, Bassi GL, Coenye T, Donelli G, Hall-Stoodley L, Hola V, Imbert C, Kirketerp-Moller K, Lebeaux D, Oliver A, Ullmann AJ, Williams C; ESCMID Study Group for Biofilms and Consulting External Expert Werner Zimmerli. ESCMID guideline for the diagnosis and treatment of biofilm infections 2014. Clin Microbiol Infect. 2015 May;21 Suppl 1:S1-25. doi: 10.1016/j.cmi.2014.10.024. Epub 2015 Jan 14. PMID 25596784
- [Background] Marsh RL, Thornton RB, Smith-Vaughan HC, Richmond P, Pizzutto SJ, Chang AB. Detection of biofilm in bronchoalveolar lavage from children with non-cystic fibrosis bronchiectasis. Pediatr Pulmonol. 2015 Mar;50(3):284-292. doi: 10.1002/ppul.23031. Epub 2014 Mar 18. PMID 24644254
- [Background] Folkesson A, Jelsbak L, Yang L, Johansen HK, Ciofu O, Hoiby N, Molin S. Adaptation of Pseudomonas aeruginosa to the cystic fibrosis airway: an evolutionary perspective. Nat Rev Microbiol. 2012 Dec;10(12):841-51. doi: 10.1038/nrmicro2907. Epub 2012 Nov 13. PMID 23147702
- [Background] Oliver A, Canton R, Campo P, Baquero F, Blazquez J. High frequency of hypermutable Pseudomonas aeruginosa in cystic fibrosis lung infection. Science. 2000 May 19;288(5469):1251-4. doi: 10.1126/science.288.5469.1251. PMID 10818002
- [Background] Kragh KN, Alhede M, Jensen PO, Moser C, Scheike T, Jacobsen CS, Seier Poulsen S, Eickhardt-Sorensen SR, Trostrup H, Christoffersen L, Hougen HP, Rickelt LF, Kuhl M, Hoiby N, Bjarnsholt T. Polymorphonuclear leukocytes restrict growth of Pseudomonas aeruginosa in the lungs of cystic fibrosis patients. Infect Immun. 2014 Nov;82(11):4477-86. doi: 10.1128/IAI.01969-14. Epub 2014 Aug 11. PMID 25114118
- [Background] Rogers GB, Zain NM, Bruce KD, Burr LD, Chen AC, Rivett DW, McGuckin MA, Serisier DJ. A novel microbiota stratification system predicts future exacerbations in bronchiectasis. Ann Am Thorac Soc. 2014 May;11(4):496-503. doi: 10.1513/AnnalsATS.201310-335OC. PMID 24592925
- [Background] Gallego M, Pomares X, Espasa M, Castaner E, Sole M, Suarez D, Monso E, Monton C. Pseudomonas aeruginosa isolates in severe chronic obstructive pulmonary disease: characterization and risk factors. BMC Pulm Med. 2014 Jun 26;14:103. doi: 10.1186/1471-2466-14-103. PMID 24964956
- [Background] Finch S, McDonnell MJ, Abo-Leyah H, Aliberti S, Chalmers JD. A Comprehensive Analysis of the Impact of Pseudomonas aeruginosa Colonization on Prognosis in Adult Bronchiectasis. Ann Am Thorac Soc. 2015 Nov;12(11):1602-11. doi: 10.1513/AnnalsATS.201506-333OC. PMID 26356317
- [Background] Costerton JW, Stewart PS, Greenberg EP. Bacterial biofilms: a common cause of persistent infections. Science. 1999 May 21;284(5418):1318-22. doi: 10.1126/science.284.5418.1318. PMID 10334980
- [Background] Langton Hewer SC, Smyth AR. Antibiotic strategies for eradicating Pseudomonas aeruginosa in people with cystic fibrosis. Cochrane Database Syst Rev. 2014 Nov 10;(11):CD004197. doi: 10.1002/14651858.CD004197.pub4. PMID 25383937
- [Background] Rutter WC, Burgess DR, Burgess DS. Increasing Incidence of Multidrug Resistance Among Cystic Fibrosis Respiratory Bacterial Isolates. Microb Drug Resist. 2017 Jan;23(1):51-55. doi: 10.1089/mdr.2016.0048. Epub 2016 Jun 21. PMID 27326758
- [Background] Martinez-Garcia MA, de la Rosa Carrillo D, Soler-Cataluna JJ, Donat-Sanz Y, Serra PC, Lerma MA, Ballestin J, Sanchez IV, Selma Ferrer MJ, Dalfo AR, Valdecillos MB. Prognostic value of bronchiectasis in patients with moderate-to-severe chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2013 Apr 15;187(8):823-31. doi: 10.1164/rccm.201208-1518OC. PMID 23392438
- [Background] Sethi S, Evans N, Grant BJ, Murphy TF. New strains of bacteria and exacerbations of chronic obstructive pulmonary disease. N Engl J Med. 2002 Aug 15;347(7):465-71. doi: 10.1056/NEJMoa012561. PMID 12181400
- [Background] Huerta A, Crisafulli E, Menendez R, Martinez R, Soler N, Guerrero M, Montull B, Torres A. Pneumonic and nonpneumonic exacerbations of COPD: inflammatory response and clinical characteristics. Chest. 2013 Oct;144(4):1134-1142. doi: 10.1378/chest.13-0488. PMID 23828375
- [Background] Domenech A, Puig C, Marti S, Santos S, Fernandez A, Calatayud L, Dorca J, Ardanuy C, Linares J. Infectious etiology of acute exacerbations in severe COPD patients. J Infect. 2013 Dec;67(6):516-23. doi: 10.1016/j.jinf.2013.09.003. Epub 2013 Sep 20. PMID 24055804
- [Background] Murphy TF, Brauer AL, Eschberger K, Lobbins P, Grove L, Cai X, Sethi S. Pseudomonas aeruginosa in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2008 Apr 15;177(8):853-60. doi: 10.1164/rccm.200709-1413OC. Epub 2008 Jan 17. PMID 18202344
- [Background] Murphy TF. Pseudomonas aeruginosa in adults with chronic obstructive pulmonary disease. Curr Opin Pulm Med. 2009 Mar;15(2):138-42. doi: 10.1097/MCP.0b013e328321861a. PMID 19532029
- [Background] Martinez-Solano L, Macia MD, Fajardo A, Oliver A, Martinez JL. Chronic Pseudomonas aeruginosa infection in chronic obstructive pulmonary disease. Clin Infect Dis. 2008 Dec 15;47(12):1526-33. doi: 10.1086/593186. PMID 18990062
- [Background] Polverino E, Goeminne PC, McDonnell MJ, Aliberti S, Marshall SE, Loebinger MR, Murris M, Canton R, Torres A, Dimakou K, De Soyza A, Hill AT, Haworth CS, Vendrell M, Ringshausen FC, Subotic D, Wilson R, Vilaro J, Stallberg B, Welte T, Rohde G, Blasi F, Elborn S, Almagro M, Timothy A, Ruddy T, Tonia T, Rigau D, Chalmers JD. European Respiratory Society guidelines for the management of adult bronchiectasis. Eur Respir J. 2017 Sep 9;50(3):1700629. doi: 10.1183/13993003.00629-2017. Print 2017 Sep. PMID 28889110
- [Background] Wang Z, Singh R, Miller BE, Tal-Singer R, Van Horn S, Tomsho L, Mackay A, Allinson JP, Webb AJ, Brookes AJ, George LM, Barker B, Kolsum U, Donnelly LE, Belchamber K, Barnes PJ, Singh D, Brightling CE, Donaldson GC, Wedzicha JA, Brown JR; COPDMAP. Sputum microbiome temporal variability and dysbiosis in chronic obstructive pulmonary disease exacerbations: an analysis of the COPDMAP study. Thorax. 2018 Apr;73(4):331-338. doi: 10.1136/thoraxjnl-2017-210741. Epub 2017 Dec 21. PMID 29269441
- [Background] Martinez-Garcia MA, Maiz L, Olveira C, Giron RM, de la Rosa D, Blanco M, Canton R, Vendrell M, Polverino E, de Gracia J, Prados C. Spanish Guidelines on the Evaluation and Diagnosis of Bronchiectasis in Adults. Arch Bronconeumol (Engl Ed). 2018 Feb;54(2):79-87. doi: 10.1016/j.arbres.2017.07.015. Epub 2017 Nov 9. English, Spanish. PMID 29128130
- [Background] Cox MJ, Turek EM, Hennessy C, Mirza GK, James PL, Coleman M, Jones A, Wilson R, Bilton D, Cookson WO, Moffatt MF, Loebinger MR. Longitudinal assessment of sputum microbiome by sequencing of the 16S rRNA gene in non-cystic fibrosis bronchiectasis patients. PLoS One. 2017 Feb 7;12(2):e0170622. doi: 10.1371/journal.pone.0170622. eCollection 2017. PMID 28170403
- [Background] Taylor SL, Woodman RJ, Chen AC, Burr LD, Gordon DL, McGuckin MA, Wesselingh S, Rogers GB. FUT2 genotype influences lung function, exacerbation frequency and airway microbiota in non-CF bronchiectasis. Thorax. 2017 Apr;72(4):304-310. doi: 10.1136/thoraxjnl-2016-208775. Epub 2016 Aug 8. PMID 27503233
- [Background] Crisafulli E, Torres A, Huerta A, Guerrero M, Gabarrus A, Gimeno A, Martinez R, Soler N, Fernandez L, Wedzicha JA, Menendez R. Predicting In-Hospital Treatment Failure (</= 7 days) in Patients with COPD Exacerbation Using Antibiotics and Systemic Steroids. COPD. 2016;13(1):82-92. doi: 10.3109/15412555.2015.1057276. Epub 2015 Oct 9. PMID 26451913
- [Background] He X, Hu W, He J, Guo L, Lux R, Shi W. Community-based interference against integration of Pseudomonas aeruginosa into human salivary microbial biofilm. Mol Oral Microbiol. 2011 Dec;26(6):337-52. doi: 10.1111/j.2041-1014.2011.00622.x. Epub 2011 Sep 13. PMID 22053962
- [Background] Brill SE, Patel AR, Singh R, Mackay AJ, Brown JS, Hurst JR. Lung function, symptoms and inflammation during exacerbations of non-cystic fibrosis bronchiectasis: a prospective observational cohort study. Respir Res. 2015 Feb 7;16(1):16. doi: 10.1186/s12931-015-0167-9. PMID 25849856
- [Background] Tacconelli E, Carrara E, Savoldi A, Harbarth S, Mendelson M, Monnet DL, Pulcini C, Kahlmeter G, Kluytmans J, Carmeli Y, Ouellette M, Outterson K, Patel J, Cavaleri M, Cox EM, Houchens CR, Grayson ML, Hansen P, Singh N, Theuretzbacher U, Magrini N; WHO Pathogens Priority List Working Group. Discovery, research, and development of new antibiotics: the WHO priority list of antibiotic-resistant bacteria and tuberculosis. Lancet Infect Dis. 2018 Mar;18(3):318-327. doi: 10.1016/S1473-3099(17)30753-3. Epub 2017 Dec 21. PMID 29276051
- [Background] Doern CD. When does 2 plus 2 equal 5? A review of antimicrobial synergy testing. J Clin Microbiol. 2014 Dec;52(12):4124-8. doi: 10.1128/JCM.01121-14. Epub 2014 Jun 11. PMID 24920779
- [Background] Natan M, Banin E. From Nano to Micro: using nanotechnology to combat microorganisms and their multidrug resistance. FEMS Microbiol Rev. 2017 May 1;41(3):302-322. doi: 10.1093/femsre/fux003. PMID 28419240
- [Background] Liu Z, Jiao Y, Wang Y, Zhou C, Zhang Z. Polysaccharides-based nanoparticles as drug delivery systems. Adv Drug Deliv Rev. 2008 Dec 14;60(15):1650-62. doi: 10.1016/j.addr.2008.09.001. Epub 2008 Sep 17. PMID 18848591
- [Background] Khan S, Tondervik A, Sletta H, Klinkenberg G, Emanuel C, Onsoyen E, Myrvold R, Howe RA, Walsh TR, Hill KE, Thomas DW. Overcoming drug resistance with alginate oligosaccharides able to potentiate the action of selected antibiotics. Antimicrob Agents Chemother. 2012 Oct;56(10):5134-41. doi: 10.1128/AAC.00525-12. Epub 2012 Jul 23. PMID 22825116
- [Background] Ahmad Z, Sharma S, Khuller GK. Inhalable alginate nanoparticles as antitubercular drug carriers against experimental tuberculosis. Int J Antimicrob Agents. 2005 Oct;26(4):298-303. doi: 10.1016/j.ijantimicag.2005.07.012. PMID 16154726
- [Derived] Fernandez-Barat L, Lopez-Aladid R, Alcaraz-Serrano V, Vazquez N, Bueno-Freire L, Pastor-Ibanez R, Lingren L, Sanz-Fraile H, Oscanoa P, Motos A, Cabrera R, Vila J, Martinez D, Otero J, Farre R, Hoiby N, Torres A. Clinical and Lung Microbiome Impact of Chronic Versus Intermittent Pseudomonas aeruginosa Infection in Bronchiectasis. Arch Bronconeumol. 2025 Nov;61(11):669-679. doi: 10.1016/j.arbres.2025.03.003. Epub 2025 Mar 18. English, Spanish. PMID 40187923